CLINICAL TRIAL: NCT05053295
Title: An Open-label, Single-arm, Single-center, Investigator-initiated Pilot Study to Investigate the Efficacy and Safety of Immuncell-LC in Combination With Nivolumab (Opdivo®) in Subjects With Advanced or Recurrent Gastric Cancer
Brief Title: Investigator-initiated Pilot Study to Investigate the Efficacy and Safety of Immuncell-LC in Combination With Nivolumab (Opdivo) in Subjects With Advanced or Recurrent Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Cho, Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2020-0356
Record Dates: First submitted 2021-09-07; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Relapsed or Advanced Gastric Adenocarcinoma; Gastro-esophageal Junction Cancer
Keywords: Immuncell-LC; Nivolumab; ILC-IIT-09; gastric adenocarcinoma,; gastro-esophageal junction cancer
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immuncell-LC/Nivolumab group (Experimental): Patients will receive nivolumab once a day at 4-week intervals and Immuncell-LC 12 times (3 treatments once a week, followed by 5 treatments every other week, and finally 4 treatments every 4 weeks).
  Interventions: Drug: autologous activated T lymphocyte

INTERVENTIONS:
Drug: autologous activated T lymphocyte — Drug: Immuncell-LC IV
  Drug: Nivolumab (Opdivo®) IV
  Other Names: Immuncell-LC (Autologous activated T lymphocyte),

SUMMARY:
This study was planned to evaluate the efficacy and safety of combination therapy of Immuncell-LC and nivolumab in patients with relapsed or advanced gastric adenocarcinoma or gastro-esophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged 19 years or above
2. Histologically and/or cytologically confirmed unresectable advanced/relapsed gastric adenocarcinoma or gastro-esophageal junction cancer that meets one of the following criteria:

   A. Confirmed relapsed or advanced gastric adenocarcinoma or gastro-esophageal junction cancer after at least two prior chemotherapies (Perioperative, neoadjuvant, and adjuvant chemotherapy are not considered as prior chemotherapies, but if the disease progression occurs during or within 6 months of completion of adjuvant chemotherapy, it is considered a prior chemotherapy).

   B. Patients who are not eligible for standard anti-cancer treatments due to contraindications, intolerance, etc. or who have no other standard treatments available for refusing the treatment may be enrolled at the judgement of the investigator regardless of the number of prior chemotherapies.
3. A measurable lesion based on RECIST v1.1 (Irradiated area will be considered measurable if PD is confirmed in the area).
4. The Eastern Cooperative Oncology Group (ECOG) performance status (PS)0-1
5. Life expectancy of at least 12 weeks
6. Confirmed adequate hematological, hepatic, renal and coagulation functions as follows:

   A. Hematological function: absolute neutrophil count (ANC) ≥ 1,500/μL, hemoglobin ≥ 9 g/dL, platelet count ≥ 100,000/μL B. Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit normal (ULN), total bilirubin ≤ 1.0 × ULN (if liver metastasis is confirmed, AST/ALT < 3 × ULN) C. Renal function: blood urine nitrogen (BUN) and serum creatinine ≤ 1.5 × ULN D. Blood coagulation:prothrombin time (PT) (international normalized ratio, INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
7. Fully understood the study information (purpose, procedure, etc.) and voluntarily provided a written consent to participate in this study.

Exclusion Criteria:

* 1) Prior treatment with any cell therapy products including but not limited to Immuncell-LC or natural killer (NK) cell therapy products

  2) Prior immuno-oncology agents such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, and anti-CTLA-4

  3) Hypersensitivity to the active ingredient or excipients of Immuncell-LC or nivolumab

  4) Unable to collect autologous blood for production of Immuncell-LC at the judgement of the investigator

  5) History of anti-cancer treatment (chemotherapy, targeted therapy [within 4 weeks for monoclonal antibody], radiation therapy, etc.) within 2 weeks prior to screening

  6) An adverse event (AE) with prior treatments that is not resolved (CTCAE grade ≤ 1 or baseline) (with the exceptions of peripheral neuropathy or alopecia that are ≥ grade 2)

  7) History of immunosuppressive drugs within 2 weeks prior to screening (with the exceptions of topical, ophthalmic, intra-articular, intranasal, or inhalational corticosteroids, or systemic corticosteroids at doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid)

  8) Administration of live vaccines, live attenuated vaccines, or inactivated vaccines within 4 weeks prior to screening

  9) The following medical history confirmed at screening: A. Confirmed diagnosis of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) which could worsen by immunotherapy B. History of an active immune disease (e.g. rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, multiple sclerosis, T cell lymphoma) with systemic treatment (disease controllers, corticosteroids, immunosuppressants, etc.) within 2 years prior to screening (Alternative therapies [e.g., thyroxine, insulin, physiologic replacement therapy with corticosteroids for adrenal or pituitary insufficiency] are not considered as systemic treatments) C. History of interstitial lung disease D. Concurrent infection or sepsis E. Evident myocardial failure or uncontrolled arterial hypertension F. Gastrointestinal perforation or fistula G. History of other malignant tumors excluding gastric adenocarcinoma/gastro-esophageal junction cancer within 5 years prior to screening (If the investigator determines that basal cell carcinoma/squamous cell carcinoma of the skin, localized prostate cancer, papillary thyroid carcinoma, or cervical carcinoma in situ is cured after successful treatment, the patients are eligible to participate even if 5 years have not passed)

  10) The following concomitant diseases at screening that may affect the safety and efficacy assessments during the study at the judgement of the investigator: A. Clinically significant pericardial effusion, pleural effusion or ascites (e.g., requiring treatment) B. Clinically significant symptoms or uncontrolled central nervous system or brain metastases or carcinomatous meningitis (except if progression is not confirmed clinically and on CT/MRI for at least 4 weeks before administration of the IP and treatment with steroids, etc. is not required for 7 days before administration of the IP after treatment of central nervous system or brain metastases.) C. Diseases that may clinically increase the risk of gastrointestinal bleeding (e.g., active diverticulitis, gastro-intestinal ulcerative disease or disease that can increase the risk of perforation) D. Active hepatitis B (HbsAg positive) or C (The patients are eligible to participate in the study even if HCV antibody is positive as long as RNA is negative, as it will be considered as a prior infection) E. Severe infections or other uncontrolled active infectious diseases requiring administration of antibiotics, antivirals, etc. that may affect the safety and efficacy assessments during the study F. Thromboembolic diseases or bleeding diatheses G. Considered ineligible to participate in the study due to concomitant disease that is uncontrolled or requires treatment (e.g., heart disease, decreased lung function, decreased kidney function, hypotension, hypertension, findings of myelosuppression, hepatitis, liver cirrhosis, history of alcohol addiction, myocardial infarction)

  11) Pregnant or breast-feeding women, or women who intend to become pregnant

  12) Received other IP or used an investigational device within 4 weeks prior to screening

  13) Ineligible or unable to participate in the study at the judgement of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on RECIST v1.1 | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months after Last Patient In)
  ORR is defined as the number of subjects with a best overall response (BOR) of complete response (CR) or partial response (PR) and expressed as a percentage of all treated participants.

SECONDARY OUTCOMES:
Overall survival (OS) | Until death, follow-up failure or study discontinuation (Up to approximately 12 months after Last Patient In)
  Overall survival is defined as the time from randomization to death due to any cause.
Progression-free survival (PFS) based on RECIST v1.1 | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months from the date the last subject was administered)
  PFS is defined as the time from the date of enrollment day to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1
Duration of response (DOR) based on RECIST v1.1 | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months from the date the last subject was administered)
  DOR is defined as the time from the earliest date of qualifying response (CR or PR) until earliest date of disease progression or death from any cause, whichever comes first. Responses are according to RECIST 1.1
Disease control rate (DCR) based on RECIST v1.1 | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months from the date the last subject was administered)
  DCR is defined as the percentage of participants in the analysis population who have CR (disappearance of all lesions), PR (≥30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters), or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD). Responses are according to RECIST 1.1
ORR based on iRECIST | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months from the date the last subject was administered)
  ORR is defined as the percentage of participants who have a best response of Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline sum diameters). Responses are according to iRECIST
PFS based on iRECIST | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months from the date the last subject was administered)
  PFS is defined as the time from the date of enrollment day to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to iRECIST
DOR based on iRECIST | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months from the date the last subject was administered)
  DOR is defined as the time from the earliest date of qualifying response (CR or PR) until earliest date of disease progression or death from any cause, whichever comes first. Responses are according to iRECIST
DCR based on iRECIST | Until disease progression, withdrawn, or initiation of subsequent chemotherapy (Up to approximately 12 months from the date the last subject was administered)
  DCR is defined as the percentage of participants in the analysis population who have CR (disappearance of all lesions), PR (≥30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters), or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD). Responses are according to iRECIST
Quality of life (QoL) assessment using the EORTC QLQ-STO22 | Until end of treatment (Up to approximately 12 months from the date the last subject was administered)
  EORTC STO-22 (European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire Gastric Module (STO = stomach) (22 items), comprising five multi-item and four single-item subscales. The multi-item subscales include questions about dysphagia (4 items), dietary restriction (5 items), pain (3 items), upper gastro-esophageal symptoms such as reflux (3 items), and emotional problems such as anxiety (3 items). The single-item subscales include questions related to four gastric cancer-specific symptoms: dry mouth, body image, hair loss, and problems with taste. Items are assessed on a 4-level numerical scale with 1= "not at all", 2= "a little", 3= "quite a bit", and 4= "very much". Scores are linearly converted and summated into a scaled score from 0 to 100, with a higher score representing a worse QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Cho, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severacen Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No